CLINICAL TRIAL: NCT00186147
Title: Bone Marrow Grafting for Leukemia and Lymphoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB-08903; P01CA049605 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Leukemia; Lymphoma; Hematologic Diseases
MeSH Terms: conditions — Leukemia; Lymphoma; Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples will be obtained from subjects undergoing transplantation or donors providing the graft.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Graft recipients and donors
  Interventions: Procedure: collection and storage of tissue samples for research

INTERVENTIONS:
Procedure: collection and storage of tissue samples for research — Tissue samples include blood draws for the donor and recipient. A bone marrow sample may be obtained from the recipient. If the recipient undergoes a tissue biopsy for clinical reasons, a small fraction may be removed for research purposes. A small fraction of the donor graft may be removed at the time of collection for research.

SUMMARY:
The purpose of this study is to obtain tissue samples for ongoing studies regarding transplant outcomes and complications.

DETAILED DESCRIPTION:
The purpose of this study is to acquire critical tissue and biological samples that can be evaluated to elucidate underlying mechanisms of disease control, transplant related complications and overall outcomes

ELIGIBILITY:
Inclusion Criteria:- All hematopoietic cell transplant recipients and donors who agree to participate

Exclusion Criteria:- Subject does not agree to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hematopoietic cell transplant recipients and donors who agree to participate
Sampling Method: Non-Probability Sample
Enrollment: 9999 (Estimated)
Dates: Start 1988-03; Primary Completion 2069-12 (Estimated); Study Completion 2069-12 (Estimated)

PRIMARY OUTCOMES:
Identify and characterize proteins and genes that may contribute to the development and progression of cancer. | blood sample is collected prior transplant, periodically during the first three months and then indefinately at follow up

CONTACTS AND LOCATIONS:
Overall Officials: David Miklos, Principal Investigator — Stanford University; Robert S Negrin, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No